CLINICAL TRIAL: NCT07051239
Title: Enhancing Waste Clearance Through Sleep Stimulation
Brief Title: Sleep Stimulation to Enhance Waste Clearance in the Brain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: University of Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HUB2025028
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Healthy; Subjective Cognitive Decline (SCD); Mild Cognitive Impairment (MCI); Alzheimer Disease (AD)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Healthy young, auditory stimulation, then sham (Experimental)
  Interventions: Other: Closed-loop acoustic stimulation
- Healthy young, sham, then auditory stimulation (Experimental)
  Interventions: Other: Closed-loop acoustic stimulation
- Healthy old, auditory stimulation, then sham (Experimental)
  Interventions: Other: Closed-loop acoustic stimulation
- Healthy old, sham then auditory stimulation (Experimental)
  Interventions: Other: Closed-loop acoustic stimulation
- Positive amyloid load group, auditory stimulation, then sham (Experimental)
  Interventions: Other: Closed-loop acoustic stimulation
- Positive amyloid load group, sham, then auditory stimulation (Experimental)
  Interventions: Other: Closed-loop acoustic stimulation

INTERVENTIONS:
Other: Closed-loop acoustic stimulation — At-home sleep will be monitored using an EEG headband. Non-awakening auditory stimuli will be delivered during non-rapid eye movement sleep (NREM), timed to the ascending phase of slow waves, using either active or control (sham) conditions.

SUMMARY:
This study aims to examine whether multi-night closed-loop auditory stimulation (CLAS) during sleep can enhance waste clearance and memory consolidation in healthy adults and older adults with subjective cognitive decline or mild cognitive impairment who exhibit elevated brain amyloid levels identified through prior clinical screening. Specifically, the study investigates whether sleep stimulation increases the clearance of plasma biomarkers related to neurodegeneration, improves the brain's waste clearance system, and supports memory consolidation. Participants will undergo five nights each of CLAS and sham (no stimulation) interventions, with a washout period in between. They will also complete clinical assessments, including MRI scans, blood sample collection, and cognitive testing, and will keep track of subjective sleep quality, sleepiness, mood, and fatigue throughout the interventions.

ELIGIBILITY:
For the positive amyloid load group:

-Participants who meet the criteria of subjective cognitive decline or mild cognitive impairment (Clinical Dementia Rating < 2; Mini-Mental State Examination ≥ 21) and brain amyloid-beta (Aβ) accumulation confirmed by CSF or amyloid-PET, the inclusion age range is 55-80 years.

For healthy groups:

-Inclusion age range is 18-80 years.

Inclusion criteria:

* Proficiency in the French language (close to native level) to complete the neuropsychological evaluation and cognitive tests.
* MRI compatibility: absence of metallic materials in the body (implants, vascular clips, certain types of orthopedic material, etc.), a pacemaker or other types of stimulators, cochlear implants, or any other electronic devices.

Exclusion criteria:

* Current or past psychiatric or neurological conditions (except for those directly associated with the patient group).
* The presence of severe untreated sleep disorders.
* The presence of irregular sleep-wake cycles (due to shiftwork or extreme chronotype).
* The presence of moderate depression or high levels of anxiety.
* Ongoing treatment with psychotropic medications (benzodiazepines, antidepressants).
* Regular or excessive consumption of alcohol or caffeinated drinks.
* Consumption of other psychoactive substances known to have an impact on the central nervous system.
* Insufficient visual or auditory acuity to complete the assessments if uncorrected. Normal hearing is required for sound stimulation to be effective.
* Claustrophobia that prevents undergoing brain imaging (MRI).
* Pregnancy or currently breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Plasma biomarkers | Blood samples will be collected the morning after each intervention phase. Interventions are separated by one week.
  Levels of plasma biomarkers associated with neurodegeneration and brain health will be compared between stimulation and sham interventions.

SECONDARY OUTCOMES:
Glymphatic function | MRI scans will be performed the morning after each intervention phase. Interventions are separated by one week.
  Magnetic resonance imaging (MRI) derived measures will serve as proxies for glymphatic function and will be compared between stimulation and sham interventions.
CLAS evoked responses | Each night of sleep during each intervention phase, whether receiving stimulation or sham.
  EEG responses locked to the acoustic stimulation will be examined (phase, amplitude, power, slow oscillations, spindle coupling) during stimulation and sham night recordings. Associations between APOE phenotype, age, amyloid accumulation, brain structure and function, baseline memory performance, sleep quality and responses to CLAS will be evaluated.
Slow wave activity (SWA) | Each night of sleep during each intervention phase, whether receiving stimulation or sham.
  EEG SWA will be assessed during NREM sleep periods from each intervention (stimulation and sham)
Sleep architecture | Each night of sleep during each intervention phase, whether receiving stimulation or sham.
  As measured with the EEG headband, macro- (e.g., duration, latency, distribution of sleep stages), and micro-architecture (slow waves, sleep spindles, rapid eye movements, arousals) differences between stimulation and sham conditions will be assessed.
Change in memory performance | Before and after each intervention period. Interventions are separated by one week.
  Performance change in declarative memory tasks (cued-recall and recognition measures) will be evaluated.
Encoding capacity | After each intervention phase. Interventions are separated by one week.
  Performance in a continuous mnemonic discrimination task (recognition and mnemonic discrimination measures) will be assessed after both stimulation and sham interventions.
Alertness and sustained attention | The PVT task will be assessed before and after each intervention phase. Interventions are separated by one week.
  Performance (reaction times, lapses) in the psychomotor vigilance task (PVT).
Subjective measures after sleep | Each morning throughout the intervention phase.
  As measured with morning questionnaires, subjective sleep quality, fatigue, sleepiness, mood, and affect, will be assessed every morning during each stimulation and sham intervention.
Resting-state functional connectivity | MRI scans will be performed the morning after each intervention phase. Interventions are separated by one week.
  Changes in resting-state functional connectivity measured with fMRI will be compared between stimulation and sham interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Strauss, MD, PhD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Hôpital Universitaire de Bruxelles, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes